CLINICAL TRIAL: NCT00376662
Title: HRT and/or Etidronate in the Prevention and Treatment of Osteoporosis and Fractures in Post-Menopausal Patients With Asthma Receiving Long-Term Oral and/or Inhaled Glucocorticoids:a Randomised Factorial Trial
Brief Title: HRT Versus Etidronate for Osteoporosis and Fractures in Asthmatics Receiving Glucocorticoids.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: British Thoracic Society (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BTS HRT and Etidronate Study
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Osteoporosis
Keywords: HRT; Etidronate; Fractures; Osteoporosis; Asthma; Glucocorticoids
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Asthma | interventions — Hormone Replacement Therapy; Etidronic Acid

INTERVENTIONS:
Drug: Hormone Replacement Therapy and Etidronate

SUMMARY:
To determine and compare the effects of Hormone replacement therapy (HRT), etidronate, HRT plus etidronate and no treatment over 5 years in the prevention and treatment of glucocorticoid-induced osteoporosis and fractures in post-menopausal women with asthma.

DETAILED DESCRIPTION:
Multicentre trial involving 13 hospitals in United Kingdom, with patients entered by 17 Consultant Chest Physicians. Consenting patients were randomised in a central office to either HRT, etidronate, HRT plus etidronate or no treatment. Information on the progress of the patients was requested by the co-ordinating office annually for 5 years after entry to the trial. Outcomes were measured as new symptomatic fractures,new or worsening morphometric fractures of the thoraco-lumbar spine and changes in bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, asthmatic outpatients under 60 years of age on long-term oral or inhaled glucocorticoid treatment for at least one year.

Exclusion Criteria:

* Hysterectomy, history of breast or endometrial cancer, undiagnosed pelvic or breast mass, untreated hypertension.

Ages: 0 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 750
Dates: Start 1992-08; Study Completion 2000-10

PRIMARY OUTCOMES:
New symptomatic fractures, new or worsening morphometric fractures of the throaco-lumbar spine, and changes in bone mineral density.

SECONDARY OUTCOMES:
Unwanted effects

CONTACTS AND LOCATIONS:
Overall Officials: Roger M Francis, MD, Study Director — School of Clinical Medical Studies University of Newcastle, UK.
Locations (2):
- United Kingdom (2):
  - Department of Chest Medicine, Llandough Hospital, Cardiff, Wales
  - Department of Chest Medicine, Llandough Hospital,, Cardiff, Wales

REFERENCES:
- [Derived] Campbell IA, Douglas JG, Francis RM, Prescott RJ, Reid DM; Research Committee of the British Thoracic Society. Hormone replacement therapy (HRT) or etidronate for osteoporosis in postmenopausal asthmatics on glucocorticoids: a randomised factorial trial. Scott Med J. 2009 Feb;54(1):21-5. doi: 10.1258/rsmsmj.54.1.21. PMID 19291931